CLINICAL TRIAL: NCT01301196
Title: An Intervention to Decrease Sedentary Behaviour in Young Adults at Risk of type2 Diabetes Mellitus - Project STAND
Brief Title: Reducing Sedentary Behaviour in Young Adults at Risk of Diabetes
Acronym: STAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loughborough University (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Stuart Biddle / Professor, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MRC 91409
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2010-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: sedentary behaviour; diabetes; structured education; 18-30 years olds; family history of T2DM or CVD; BMI ≥ 25 (≥23 for south Asians)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Behaviour change (Experimental): Attendance at 3-h workshop
  Interventions: Behavioral: Educational workshop

INTERVENTIONS:
Behavioral: Educational workshop — 3h attendance at educational workshop plus self-monitoring

SUMMARY:
Excessive periods of time spent sitting may be a risk factor for diabetes. Current lifestyles encourage large amounts of sitting (sedentary behaviour) through increasing car use, computers, and appealing screen-based home entertainment systems. Methods to help change such behaviours are now needed, particularly for those with a high risk of developing a chronic disease, such as diabetes. The investigators propose to decrease sedentary behaviour in a multi-ethnic group of young adults at risk of diabetes through an educational intervention (attending a workshop and having prompts). If successful, this could have significant public health benefits given the widespread nature of sedentary behaviour.

DETAILED DESCRIPTION:
The rising prevalence of obesity and sedentary behaviour has lead to an epidemic of Type 2 Diabetes (T2DM). As the health and economic costs of T2DM continue to increase, there is an urgent need for an effective lifestyle intervention to prevent the development of T2DM. Our group have previously developed successful structured education programmes: DESMOND improved lifestyle, depression, illness beliefs, weight and CV risk in adults with T2DM; PREPARE increased activity levels and reduced 2 hour glucose values in people with pre-diabetes. Project STAND will assess the effect of theory driven structured education, facilitated using automated technology, on sedentary behaviour and health outcomes in young adults at risk of T2DM. Participants will be randomised to a control (C) or intervention (I) group, the latter given structured education, based on the PREPARE and DESMOND programmes, with the aim of reducing sedentary behaviour. The structured education programme will incorporate movement technology to facilitate participant feedback and self-monitoring.This will be the first UK trial to address sedentary behaviour change in a population of younger adults at risk of T2DM. Our results will provide a platform for the development of a range of future multidisciplinary interventions in this rapidly expanding high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-30 years old
* family history of T2DM or CVD (first degree relative)
* BMI ≥ 25 (≥ 23 for south Asians)

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 189 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Sedentary behaviour | 12 months
  Sedentary behaviour (time < 100 counts/min as assessed by 1-week accelerometry, using the new Actigraph GT3X) at 12 months

SECONDARY OUTCOMES:
Biomarkers | 12 months
  Fasting and 2h glucose, blood lipid profile, insulin, HbA1c, hsCRP, TNFα, IL-6, and IL-6
Screen time | 12 months
  self-reported screen-time (TV, computers, games)
Self-reported behaviour | 12 months
  Time in motorised transport, physical activity (accelerometer and IPAQ questionnaire)
Biological measures | 12 months
  Body weight, waist circumference, blood pressure
Psychosocial indicators | 12 months
  Illness perceptions (brief IPQ), efficacy beliefs

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester, Leicester, Leics, United Kingdom